CLINICAL TRIAL: NCT03546114
Title: Does Gender Matter? Patient Preference in an Italian Osteopathic Clinical Setting
Status: Completed | Type: Observational
Sponsor: Istituto Superiore di Osteopatia di Milano (Other)
Responsible Party: Principal Investigator, Viviana Pisa, PhD, Istituto Superiore di Osteopatia di Milano
Other Study IDs: 052018
Record Dates: First submitted 2018-05-21; First posted 2018-06-06 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Gender Role
Keywords: Gender; Sex and gender; Patient preference; Osteopathic medicine
MeSH Terms: conditions — Coitus; Patient Preference

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients referring to an osteopathic clinic - CMO, Milan: Adults, age>18 years, first visit at osteopathic clinic (Centro di Medicina Osteopatica)
  Interventions: Other: Gender Questionnaire

INTERVENTIONS:
Other: Gender Questionnaire — 13-items questionnaire including demographics questions (gender, age, education; naive to osteopathic treatment or not; general gender preferences; specific gender preference in case of low back pain, neck pain, gastrointestinal disorders, musculoskeletal disorders of upper and lower limbs pain; headache; urogenital disorders

SUMMARY:
This study evaluates patients preference for the gender of their osteopath. All patients referring to an Italian private osteopathic clinic will receive a proper questionnaire before knowing the gender of their designed osteopath.

DETAILED DESCRIPTION:
Several previous studies have shown that clinical contextual factors, such as patients preferences, play an important role in the patient-physical relationship, with resulting consequences on clinical outcomes.

The interaction between the gender of both patient and physician is often impacted by existing stereotypes.

Patient preference for specific physician gender has been investigated in scientific literature.

However the are no studies that analyzed the role of gender in osteopathic medicine.

ELIGIBILITY:
Inclusion Criteria: first visit at the osteopathic clinic (Centro di Medicina Osteopatica) Milan

Exclusion Criteria: non-Italian speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients referring to Centro di Medicina Osteopatica for the first visit.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Gender questionnaire (Self-reported 13-items questionnaire) | 1 day
  * Patient's gender?
  * Patient's age?
  * Educational level? (middle school, high school, BSc, MSc, PhD)
  * Naive to osteopathic treatment? (yes/no)
  * Only if the answer of question 5 is yes, which was the osteopath's gender at your first osteopathic consultation?
  * Which would be your favorite osteopath's gender?
  * Which would be your favorite osteopath's gender if you had low back pain?
  * Which would be your favorite osteopath's gender if you had neck pain?
  * Which would be your favorite osteopath's gender if you had gastrointestinal disorders?
  * Which would be your favorite osteopath's gender if you had upper limb pain?
  * Which would be your favorite osteopath's gender if you had lower limb pain?
  * Which would be your favorite osteopath's gender if you had headache?
  * Which would be your favorite osteopath's gender if you had urogenital disorders? Questions 7-13: Choose among: female, male, no preference

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ratti, MSc, Principal Investigator — Istituto Superiore di Osteopatia (ISO)
Locations (1):
- Istituto Superiore di Osteopatia, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Background] Abghari MS, Takemoto R, Sadiq A, Karia R, Phillips D, Egol KA. Patient perceptions and preferences when choosing an orthopaedic surgeon. Iowa Orthop J. 2014;34:204-8. PMID 25328483
- [Background] Alvarez Bustins G, Lopez Plaza PV, Carvajal SR. Profile of osteopathic practice in Spain: results from a standardized data collection study. BMC Complement Altern Med. 2018 Apr 11;18(1):129. doi: 10.1186/s12906-018-2190-0. PMID 29642901
- [Background] Amir H, Beri A, Yechiely R, Amir Levy Y, Shimonov M, Groutz A. Do Urology Male Patients Prefer Same-Gender Urologist? Am J Mens Health. 2018 Sep;12(5):1379-1383. doi: 10.1177/1557988316650886. Epub 2016 May 24. PMID 27222116
- [Background] Amodio DM. The neuroscience of prejudice and stereotyping. Nat Rev Neurosci. 2014 Oct;15(10):670-82. doi: 10.1038/nrn3800. Epub 2014 Sep 4. PMID 25186236
- [Background] Balayla J. Male physicians treating Female patients: Issues, Controversies and Gynecology. Mcgill J Med. 2011 Jun;13(1):72. No abstract available. PMID 22399872
- [Background] Bishop FL, Massey Y, Yardley L, Lewith GT. How patients choose acupuncturists: a mixed-methods project. J Altern Complement Med. 2011 Jan;17(1):19-25. doi: 10.1089/acm.2010.0061. Epub 2011 Jan 16. PMID 21235412
- [Background] Bishop FL, Bradbury K, Hj Jeludin NN, Massey Y, Lewith GT. How patients choose osteopaths: a mixed methods study. Complement Ther Med. 2013 Feb;21(1):50-7. doi: 10.1016/j.ctim.2012.10.003. Epub 2012 Nov 15. PMID 23374205
- [Background] Blanch-Hartigan D, Hall JA, Roter DL, Frankel RM. Gender bias in patients' perceptions of patient-centered behaviors. Patient Educ Couns. 2010 Sep;80(3):315-20. doi: 10.1016/j.pec.2010.06.014. Epub 2010 Jul 17. PMID 20638813
- [Background] Burke SR, Myers R, Zhang AL. A profile of osteopathic practice in Australia 2010-2011: a cross sectional survey. BMC Musculoskelet Disord. 2013 Aug 1;14:227. doi: 10.1186/1471-2474-14-227. PMID 23915239
- [Background] Cerritelli F, van Dun PLS, Esteves JE, Consorti G, Sciomachen P, Lacorte E, Vanacore N; OPERA-IT Group. The Italian Osteopathic Practitioners Estimates and RAtes (OPERA) study: A cross sectional survey. PLoS One. 2019 Jan 25;14(1):e0211353. doi: 10.1371/journal.pone.0211353. eCollection 2019. PMID 30682169
- [Background] Cerritelli F, Verzella M, Barlafante G. Quality of life in patients referring to private osteopathic clinical practice: a prospective observational study. Complement Ther Med. 2014 Aug;22(4):625-31. doi: 10.1016/j.ctim.2014.05.007. Epub 2014 May 24. PMID 25146065
- [Background] Cil TD, Easson AM. The role of gender in patient preference for breast surgical care - a comment on equality. Isr J Health Policy Res. 2018 Jul 9;7(1):37. doi: 10.1186/s13584-018-0231-2. PMID 29983118
- [Background] Consorti F, Mancuso R, Piccolo A, Consorti G, Zurlo J. Evaluation of the acceptability of Peer Physical Examination (PPE) in medical and osteopathic students: a cross sectional survey. BMC Med Educ. 2013 Aug 22;13:111. doi: 10.1186/1472-6920-13-111. PMID 23968312
- [Background] Furnham A, Petrides KV, Temple J. Patient preferences for medical doctors. Br J Health Psychol. 2006 Sep;11(Pt 3):439-49. doi: 10.1348/135910705X67529. PMID 16870054
- [Background] Grinberg M, Lopes AS. Feminization of medicine. Arq Bras Cardiol. 2013 Sep;101(3):283. doi: 10.5935/abc.20130175. No abstract available. PMID 24061755
- [Background] Groutz A, Amir H, Caspi R, Sharon E, Levy YA, Shimonov M. Do women prefer a female breast surgeon? Isr J Health Policy Res. 2016 Dec 1;5:35. doi: 10.1186/s13584-016-0094-3. eCollection 2016. PMID 27980717
- [Background] Hall JA, Roter DL. Do patients talk differently to male and female physicians? A meta-analytic review. Patient Educ Couns. 2002 Dec;48(3):217-24. doi: 10.1016/s0738-3991(02)00174-x. PMID 12477606
- [Background] Janssen SM, Lagro-Janssen AL. Physician's gender, communication style, patient preferences and patient satisfaction in gynecology and obstetrics: a systematic review. Patient Educ Couns. 2012 Nov;89(2):221-6. doi: 10.1016/j.pec.2012.06.034. Epub 2012 Jul 21. PMID 22819711
- [Background] Johnson SM, Kurtz ME. Osteopathic manipulative treatment techniques preferred by contemporary osteopathic physicians. J Am Osteopath Assoc. 2003 May;103(5):219-24. PMID 12776762
- [Background] Myers SS, Phillips RS, Davis RB, Cherkin DC, Legedza A, Kaptchuk TJ, Hrbek A, Buring JE, Post D, Connelly MT, Eisenberg DM. Patient expectations as predictors of outcome in patients with acute low back pain. J Gen Intern Med. 2008 Feb;23(2):148-53. doi: 10.1007/s11606-007-0460-5. Epub 2007 Dec 8. PMID 18066631
- [Background] Lahat A, Assouline-Dayan Y, Katz LH, Fidder HH. The preference for an endoscopist specific sex: a link between ethnic origin, religious belief, socioeconomic status, and procedure type. Patient Prefer Adherence. 2013 Sep 9;7:897-903. doi: 10.2147/PPA.S48468. eCollection 2013. PMID 24043933
- [Background] McCall B. What does the GDPR mean for the medical community? Lancet. 2018 Mar 31;391(10127):1249-1250. doi: 10.1016/S0140-6736(18)30739-6. No abstract available. PMID 29619949
- [Background] Morin C, Aubin A. Primary reasons for osteopathic consultation: a prospective survey in Quebec. PLoS One. 2014 Sep 3;9(9):e106259. doi: 10.1371/journal.pone.0106259. eCollection 2014. PMID 25184204
- [Background] Nolen HA, Moore JX, Rodgers JB, Wang HE, Walter LA. Patient Preference for Physician Gender in the Emergency Department. Yale J Biol Med. 2016 Jun 27;89(2):131-42. eCollection 2016 Jun. PMID 27354840
- [Background] Olsson M, Martiny SE. Does Exposure to Counterstereotypical Role Models Influence Girls' and Women's Gender Stereotypes and Career Choices? A Review of Social Psychological Research. Front Psychol. 2018 Dec 7;9:2264. doi: 10.3389/fpsyg.2018.02264. eCollection 2018. PMID 30581398
- [Background] Rasky E, Waxenegger A, Groth S, Stolz E, Schenouda M, Berzlanovich A. Sex and gender matters : A sex-specific analysis of original articles published in the Wiener klinische Wochenschrift between 2013 and 2015. Wien Klin Wochenschr. 2017 Nov;129(21-22):781-785. doi: 10.1007/s00508-017-1280-1. Epub 2017 Oct 17. PMID 29043442
- [Background] Rossettini G, Carlino E, Testa M. Clinical relevance of contextual factors as triggers of placebo and nocebo effects in musculoskeletal pain. BMC Musculoskelet Disord. 2018 Jan 22;19(1):27. doi: 10.1186/s12891-018-1943-8. PMID 29357856
- [Background] Roter DL, Hall JA. Physician gender and patient-centered communication: a critical review of empirical research. Annu Rev Public Health. 2004;25:497-519. doi: 10.1146/annurev.publhealth.25.101802.123134. PMID 15015932
- [Background] Roter DL, Hall JA, Aoki Y. Physician gender effects in medical communication: a meta-analytic review. JAMA. 2002 Aug 14;288(6):756-64. doi: 10.1001/jama.288.6.756. PMID 12169083
- [Background] Shan G, Gerstenberger S. Fisher's exact approach for post hoc analysis of a chi-squared test. PLoS One. 2017 Dec 20;12(12):e0188709. doi: 10.1371/journal.pone.0188709. eCollection 2017. PMID 29261690
- [Background] Shin DW, Roter DL, Roh YK, Hahm SK, Cho B, Park HK; Board Certification Committee of The Korean Academy of Family Medicine. Physician gender and patient centered communication: the moderating effect of psychosocial and biomedical case characteristics. Patient Educ Couns. 2015 Jan;98(1):55-60. doi: 10.1016/j.pec.2014.10.008. Epub 2014 Oct 23. PMID 25457177
- [Background] Sandhu H, Adams A, Singleton L, Clark-Carter D, Kidd J. The impact of gender dyads on doctor-patient communication: a systematic review. Patient Educ Couns. 2009 Sep;76(3):348-55. doi: 10.1016/j.pec.2009.07.010. Epub 2009 Aug 3. PMID 19647969
- [Background] Sjostrom O, Holst D. Validity of a questionnaire survey: response patterns in different subgroups and the effect of social desirability. Acta Odontol Scand. 2002 Jun;60(3):136-40. doi: 10.1080/000163502753740133. PMID 12166905
- [Background] Stenberg G, Fjellman-Wiklund A, Ahlgren C. "Getting confirmation": gender in expectations and experiences of healthcare for neck or back patients. J Rehabil Med. 2012 Feb;44(2):163-71. doi: 10.2340/16501977-0912. PMID 22234575
- [Background] Street RL Jr. Gender differences in health care provider-patient communication: are they due to style, stereotypes, or accommodation? Patient Educ Couns. 2002 Dec;48(3):201-6. doi: 10.1016/s0738-3991(02)00171-4. PMID 12477604
- [Background] Testa M, Rossettini G. Enhance placebo, avoid nocebo: How contextual factors affect physiotherapy outcomes. Man Ther. 2016 Aug;24:65-74. doi: 10.1016/j.math.2016.04.006. Epub 2016 Apr 20. PMID 27133031
- [Background] Petkovic J, Trawin J, Dewidar O, Yoganathan M, Tugwell P, Welch V. Sex/gender reporting and analysis in Campbell and Cochrane systematic reviews: a cross-sectional methods study. Syst Rev. 2018 Aug 2;7(1):113. doi: 10.1186/s13643-018-0778-6. PMID 30068380
- [Background] Varadarajulu S, Petruff C, Ramsey WH. Patient preferences for gender of endoscopists. Gastrointest Endosc. 2002 Aug;56(2):170-3. doi: 10.1016/s0016-5107(02)70173-9. PMID 12145592
- [Background] Vieder JN, Krafchick MA, Kovach AC, Galluzzi KE. Physician-patient interaction: what do elders want? J Am Osteopath Assoc. 2002 Feb;102(2):73-8. PMID 11866395
- [Background] Wang MT, Degol JL. Gender Gap in Science, Technology, Engineering, and Mathematics (STEM): Current Knowledge, Implications for Practice, Policy, and Future Directions. Educ Psychol Rev. 2017 Mar;29(1):119-140. doi: 10.1007/s10648-015-9355-x. Epub 2016 Jan 13. PMID 28458499
- [Background] Barrett LF, Bliss-Moreau E. She's emotional. He's having a bad day: attributional explanations for emotion stereotypes. Emotion. 2009 Oct;9(5):649-58. doi: 10.1037/a0016821. PMID 19803587
- [Background] Carey TS, Motyka TM, Garrett JM, Keller RB. Do osteopathic physicians differ in patient interaction from allopathic physicians? An empirically derived approach. J Am Osteopath Assoc. 2003 Jul;103(7):313-8. PMID 12884943
- [Background] Chur-Hansen A. Preferences for female and male nurses: the role of age, gender and previous experience --year 2000 compared with 1984. J Adv Nurs. 2002 Jan;37(2):192-8. doi: 10.1046/j.1365-2648.2002.02079.x. PMID 11851787
- [Background] Ino T, Nakai R, Azuma T, Kimura T, Fukuyama H. Gender differences in brain activation during encoding and recognition of male and female faces. Brain Imaging Behav. 2010 Mar;4(1):55-67. doi: 10.1007/s11682-009-9085-0. PMID 20503114
- [Background] Kret ME, De Gelder B. A review on sex differences in processing emotional signals. Neuropsychologia. 2012 Jun;50(7):1211-21. doi: 10.1016/j.neuropsychologia.2011.12.022. Epub 2012 Jan 8. PMID 22245006
- [Background] LaFrance M, Hecht MA, Paluck EL. The contingent smile: a meta-analysis of sex differences in smiling. Psychol Bull. 2003 Mar;129(2):305-34. doi: 10.1037/0033-2909.129.2.305. PMID 12696842
- [Background] Nijs J, Roussel N, Paul van Wilgen C, Koke A, Smeets R. Thinking beyond muscles and joints: therapists' and patients' attitudes and beliefs regarding chronic musculoskeletal pain are key to applying effective treatment. Man Ther. 2013 Apr;18(2):96-102. doi: 10.1016/j.math.2012.11.001. Epub 2012 Dec 28. PMID 23273516
- [Background] Rizk DE, El-Zubeir MA, Al-Dhaheri AM, Al-Mansouri FR, Al-Jenaibi HS. Determinants of women's choice of their obstetrician and gynecologist provider in the UAE. Acta Obstet Gynecol Scand. 2005 Jan;84(1):48-53. doi: 10.1111/j.0001-6349.2005.00705.x. PMID 15603567
- [Background] Tourangeau R, Yan T. Sensitive questions in surveys. Psychol Bull. 2007 Sep;133(5):859-83. doi: 10.1037/0033-2909.133.5.859. PMID 17723033